CLINICAL TRIAL: NCT03983395
Title: A Phase 1/2, Open-Label, Dose-Escalation Study of ISB 1302 in Subjects With HER2-Positive Metastatic Breast Cancer
Brief Title: Study of ISB 1302 (CD3 Bispecific Ab) in HER2-positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated during Part 1 (dose escalation), and Part 2 (expansion) of the study was not initiated. This study was voluntarily terminated due to a business decision not to proceed with the ISB 1302 asset, and not due to any safety issue.
Sponsor: Ichnos Sciences SA (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISB 1302-103; IND Number 131316 (Other: FDA)
Record Dates: First submitted 2019-05-31; First posted 2019-06-12 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; GBR 1302; HER2; HER2 x CD3 bispecific antibody; ISB 1302 (CD3 Bispecific Ab) in HER2-positive Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Cohort 101 - ISB 1302 250 ng/kg (Experimental): Cohort 101, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. Dose on D1, D8, D15, D22 is 250 ng/kg
  Interventions: Biological: ISB 1302 250 ng/kg
- Part 1: Cohort 201 - ISB 1302 325 ng/kg (Experimental): Cohort 201, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. Dose on D1, D8, D15, D22 is 325 ng/kg
  Interventions: Biological: ISB 1302 325 ng/kg
- Part 1:Cohort 301- ISB 1302 325 ng/kg-D1;425 ng/kg -D8,D15,D22 (Experimental): Cohort 301, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of GBR 1302 is 325 ng/kg on D1 and 425 ng/kg on D8, D15, D22
  Interventions: Biological: ISB 1302 325 ng/kg-D1;425 ng/kg -D8,D15,D22
- Part 1:Cohort 401- ISB 1302 325 ng/kg-D1;550 ng/kg -D8,D15,D22 (Experimental): Cohort 401, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, D15, D22
  Interventions: Biological: ISB 1302 325 ng/kg-D1;550 ng/kg -D8,D15,D22
- Part1Cohort501-ISB1302 325ng/kgD1;550 ng/kg D8;700 ng/kgD15,22 (Experimental): Cohort 501, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, and 700 ng/kg on D15, D22
  Interventions: Biological: ISB 1302 325ng/kgD1;550 ng/kg D8;700 ng/kgD15,22
- Part1Cohort601-ISB1302 325ng/kgD1;550 ng/kg D8;900 ng/kgD15,22 (Experimental): Cohort 601, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, and 900 ng/kg on D15, D22
  Interventions: Biological: ISB 1302 325ng/kg D1;550 ng/kg D8;900 ng/kg D15,22
- Part 1 Cohort 701- ISB 1302 escalating doses,1200 ng/kg D15,22 (Experimental): Cohort 701, subjects will be administered ISB 1302 by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 700 ng/kg on D8, and 1200 ng/kg on D15, D22
  Interventions: Biological: ISB 1302 escalating doses,1200 ng/kg D15,22
- Part 2 (Dose Expansion) -ISB 1302 at the MTD and/or RP2D dose (Experimental): Subjects treated with ISB 1302 at the MTD and/or RP2D dose in separate groups in the Q1W and/or the Q2W dose regimen.
  Interventions: Biological: ISB 1302 at the MTD and/or RP2D dose

INTERVENTIONS:
Biological: ISB 1302 250 ng/kg — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. Dose on D1, D8, D15, D22 is 250 ng/kg
  Arms: Part 1: Cohort 101 - ISB 1302 250 ng/kg
Biological: ISB 1302 325 ng/kg — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at dose levels. Dose on D1, D8, D15, D22 is 325 ng/kg
  Arms: Part 1: Cohort 201 - ISB 1302 325 ng/kg
Biological: ISB 1302 325 ng/kg-D1;425 ng/kg -D8,D15,D22 — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 425 ng/kg on D8, D15, D22
  Arms: Part 1:Cohort 301- ISB 1302 325 ng/kg-D1;425 ng/kg -D8,D15,D22
Biological: ISB 1302 325 ng/kg-D1;550 ng/kg -D8,D15,D22 — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, D15, D22
  Arms: Part 1:Cohort 401- ISB 1302 325 ng/kg-D1;550 ng/kg -D8,D15,D22
Biological: ISB 1302 325ng/kgD1;550 ng/kg D8;700 ng/kgD15,22 — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, and 700 ng/kg on D15, D22
  Arms: Part1Cohort501-ISB1302 325ng/kgD1;550 ng/kg D8;700 ng/kgD15,22
Biological: ISB 1302 325ng/kg D1;550 ng/kg D8;900 ng/kg D15,22 — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 550 ng/kg on D8, and 900 ng/kg on D15, D22
  Arms: Part1Cohort601-ISB1302 325ng/kgD1;550 ng/kg D8;900 ng/kgD15,22
Biological: ISB 1302 escalating doses,1200 ng/kg D15,22 — ISB 1302 is administered by intravenous (IV) infusion on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle at escalating dose levels. Dose of ISB 1302 is 325 ng/kg on D1 and 700 ng/kg on D8, and 1200 ng/kg on D15, D22
  Arms: Part 1 Cohort 701- ISB 1302 escalating doses,1200 ng/kg D15,22
Biological: ISB 1302 at the MTD and/or RP2D dose — ISB 1302 at the MTD and/or RP2D dose in separate groups in the Q1W and/or the Q2W dose regimen.
  Arms: Part 2 (Dose Expansion) -ISB 1302 at the MTD and/or RP2D dose

SUMMARY:
The purpose of this study is to determine the safety profile, maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of single agent ISB1302 in subjects with HER2-positive metastatic breast cancer who have been treated with all known therapies known to confer clinical benefit.

DETAILED DESCRIPTION:
To determine the safety profile, maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of single agent ISB 1302 in subjects with HER2-positive metastatic breast cancer who have been treated with all known therapies known to confer clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Females with HER2-positive [IHC 2 +, with FISH confirmation] or 3+ [IHC or FISH] metastatic breast cancer that has progressed on last therapy. No more than 4 lines of therapy in metastatic setting (of which no more than 2 lines should be anti-HER2 antibody-based therapy).
* Measurable disease, defined as per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG ) performance-status score of 2 or less
* Adequate bone marrow, renal, and liver function.
* Recovered from any previous surgery and no history of major surgery within the last 28 days prior to start of study drug
* Must be willing to undergo pre-treatment and on-treatment biopsies in Part 1 and Part 2.

Exclusion Criteria:

* Any suspected or proven immunocompromised state, or infections, such as history of positive human immunodeficiency virus (HIV), known active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Any history or evidence of clinically significant cardiovascular disease.
* Evidence of clinically significant cardiovascular and respiratory conditions
* Previous antineoplastic treatment with immune checkpoint regulator or comparable immunotherapy within 8 weeks of starting study drug.
* Chemotherapy, radiotherapy, molecular-targeted therapy, or biological therapies (including HER2-directed therapies) within 4 weeks of starting study drug
* Hormone therapy within 2 weeks of starting study medications.
* Diagnosed with another malignancy that requires active therapy
* Brain metastases that require directed therapy.
* Has not recovered from any therapy related toxicities from previous treatments.
* Use of any investigational drug within 4 weeks from the start of study drug.
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study drug or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
MTD: Number of DLTs (dose limiting toxicities) during the first 28 days after the first administrations of study drug (i.e. Cycle 1) in each cohort. | 28 days
  MTD: Number of DLTs (dose limiting toxicities) during the first 28 days after the first administrations of study drug (i.e. Cycle 1) in each cohort.
RP2D: Incidence and severity of AEs, AESI, and SAEs, including but not limited to laboratory values, PK and biomarkers. | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  RP2D: Incidence and severity of AEs, AESI, and SAEs, including but not limited to laboratory values, PK and biomarkers.
Anti-tumor Activity of ISB 1302 administered Q1W (Part 2) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Tumor Response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) (Part 2)

SECONDARY OUTCOMES:
Incidence, nature, and intensity of AEs according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Incidence, nature, and intensity of AEs according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Antitumor activity of ISB 1302 administered Q1W (Part 1) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Tumor Response per RECIST v1.1.
Additional preliminary anti-tumor clinical activity of ISB 1302 administered (Part 2) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Tumor Response per RECIST v1.1
Pharmacokinetics of ISB 1302 administered Q1W (Part 1 and Part 2) -Cmax | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  PK parameter: Cmax - maximum observed serum concentration is estimated
Pharmacokinetics of ISB 1302 administered Q1W (Part 1 and Part 2)-tmax | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  PK parameter: tmax - time at which Cmax is observed
Pharmacokinetics of ISB 1302 administered Q1W (Part 1 and Part 2) -AUC0-tau | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  PK parameter: AUC0-tau - Area under the serum concentration-time curve over a dosing interval is estimated.
Pharmacokinetics of ISB 1302 administered Q1W (Part 1 and Part 2) - AUC0-t | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  PK parameter: AUC0-t - Area under the serum concentration-time curve over the time interval from zero to last quantifiable concentration is estimated.
Immunogenicity of ISB 1302 administered Q1W (Part 1 and Part 2) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Percent incidence of antidrug antibodies (ADA) formation assessed from baseline until end of treatment (EOT)
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) - levels of pharmacodynamic cytokines- IL-2 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Levels of cytokines, including IL-2 will be measured in peripheral blood as part of the pharmacodynamics and safety assessment to monitor for any signs of cytokine release syndrome.
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) - levels of pharmacodynamic cytokines- IL-6 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Levels of cytokines, including IL-6 will be measured in peripheral blood as part of the pharmacodynamics and safety assessment to monitor for any signs of cytokine release syndrome.
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) - levels of pharmacodynamic cytokines- IL-10 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Levels of cytokines, including IL-10 will be measured in peripheral blood as part of the pharmacodynamics and safety assessment to monitor for any signs of cytokine release syndrome.
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) - levels of pharmacodynamic cytokines- IFN-γ | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Levels of cytokines, including IFN-γ will be measured in peripheral blood as part of the pharmacodynamics and safety assessment to monitor for any signs of cytokine release syndrome.
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) - levels of pharmacodynamic cytokines- TNF-α | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Levels of cytokines, including TNF-α, will be measured in peripheral blood as part of the pharmacodynamics and safety assessment to monitor for any signs of cytokine release syndrome.
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers -CD3 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD3 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers -CD4 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD4 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers -CD8 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD8 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers -CD25 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD25 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers -CD69 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD69 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Pharmacodynamic Cellular Biomarkers - CD127 | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Cellular biomarkers to be analyzed include CD127 will be assessed by fluorescence activated cell sorting (FACS) analysis of peripheral blood leucocytes as surrogate markers for ISB 1302 activity
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include T cells | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include T cells
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include tumor microenvironment markers | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include tumor microenvironment markers
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include apoptotic markers | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include apoptotic markers
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include Tumor Mutational Burden (TMB) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include Tumor Mutational Burden (TMB)
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include Epigenetic evaluation of Tregs | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include Epigenetic evaluation of Tregs
Exploratory: Pharmacodynamic biomarkers of ISB 1302 (Part 1 and Part 2) -Tumor tissue biopsy -Analyses of the tumor tissue include Epigenetic evaluation of T helper cells | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Descriptive statistics for pharmacodynamic biomarker assessments such as Tumor tissue biopsy - Analyses of the tumor tissue include Epigenetic evaluation of T helper cells
Exploratory: Duration of treatment (Part 1 and Part 2) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Tumor response per RECIST v1.1 and iRECIST
Exploratory: Time to disease progression (Part 1 and Part 2) | Treatment cycles of 28 days, treatment cycles may continue, if there is clinical benefit, until disease progression, unacceptable toxicity, withdrawal, or end of study or cycles may continue beyond disease progression, treatment cycles for up to 6 months
  Tumor Response per RECIST v1.1 and iRECIST

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Ichnos Investigational Site 1, Gilbert, Arizona
  - Ichnos Investigational Site 5, Los Angeles, California
  - Ichnos Investigational Site 4, Louisville, Kentucky
  - Ichnos Investigational Site 2, Detroit, Michigan
  - Ichnos Investigational Site 3, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No